CLINICAL TRIAL: NCT03253237
Title: Continuous Glucose Monitoring in Patients With Diabetes Mellitus Type 2 in Primary Care
Brief Title: Primary Care - Continuous Glucose Monitoring
Acronym: PC-COSMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zagreb (Other)
Collaborators: Association of teachers in general practice / family medicine (Unknown)
Responsible Party: Principal Investigator, Valerija Bralic Lang, Valerija Bralic Lang, MD, FP, PhD, University of Zagreb
Other Study IDs: DNOOM1072014
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus; Continuous Glucose Monitoring
Keywords: Glycemic variability; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: continuous glucose monitoring (CGM) — A CGM device is to be set and take of by the GP. Before the study start all GPs will have a short education on CGM device by the diabetologist who use CGM on a daily base. Study period is seven days and includes screening before study entry and two visits. On Day 1, after screening and signing the informed consent, the CGM device is applied. Patient is instructed to keep a 7 day diary with four daily standard home blood glucose monitoring (SHBGM) along with the data on eating, physical exercise, drugs. Bayer's Contour® glucometer is used for the SHBGM. On Day 7, CGM device is took of and the data from iPro2 is uploaded to PC. At the end, each patient fill a short query on satisfaction while wearing CGM.
  Other Names: iPro™2 Medtronic

SUMMARY:
Introduction and objective: The key to optimal diabetes management is tight glucose control. Hemoglobin A1c is the gold standard to assess glycemic control but in cases of unrecognized hypoglycemia, confusing nighttime events or in cases of large variations in blood glucose, a haemoglobin A1c can not detect specific movement of blood glucose. Continuous glucose monitoring (CGM) provides informations of glucose levels in a real-time format and may be helpful for making the personalized therapy decisions desired in the era of precision medicine. Our aim is to analyse the benefit of tracking patterns of glucose values by using continuous glucose monitoring (CGM) in patients with T2DM in family medicine office.

DETAILED DESCRIPTION:
STUDY DESIGN: An observational, multicenter, cross-sectional study. A total of 20 GPs from four Croatian regions will recruit up to five subjects of both sexes from August 2017 till the end of September 2017, diagnosed with type 2 diabetes mellitus at least one year prior to study entry, aged ≥40 years, with no insulin in therapy and with clinical suspicion of hypoglycemia or with disproportion in actual glycemia na haemoglobin A1c findings. Sociodemographic, laboratory (HbA1c, fasting and postprandial glucose, total cholesterol, high density cholesterol, low density cholesterol, triglyceride and serum creatinine) and habits data will be collected. SETTING: Totally 100 of patients will be included. At primary care office each patient wear the device (iPro™2 Medtronic) subcutaneously for up to 7-days and return it to the office for download. Patients do not receive glucose alerts and only see the CGM data after it's been analyzed by the healthcare professional. A CGM device is to be set and take of by the GP. Before the study start all GPs will have a short education on CGM device by the diabetologist who use CGM on a daily base. Study period is seven days and includes screening before study entry and two visits. On Day 1, after screening and signing the informed consent, the CGM device is applied. Patient is instructed to keep a 7 day diary with four daily standard home blood glucose monitoring (SHBGM) along with the data on eating, physical exercise, drugs. Bayer's Contour® glucometer is used for the SHBGM. On Day 7, CGM device is took of and the data from iPro2 is uploaded to PC. At the end, each patient fill a short query on satisfaction while wearing CGM.

ELIGIBILITY:
Inclusion Criteria:

* T2DM diagnosed at least one year prior to study entry
* no insulin in therapy
* patients' ability to understand and answer the questionnaire by themselves
* signed informed consent

Exclusion Criteria:

* known coagulopathy
* oral anticoagulants in therapy
* skin disease that enables continuous glucose monitor device application
* febrile illness
* patient's inability to physically visit a general practitioners office
* patient's inability to answer the questionnaire by themselves

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Totally 100 of patients with type 2 diabetes mellitus diagnosed at least one year prior to study entry, aged ≥40 years, both sexes, treated in primary care, with no isulin in therapy and with clinical suspicion of hypoglycemia or with disproprtion in actual glycemia na haemoglobin A1c findings will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-10-07 (Estimated)

PRIMARY OUTCOMES:
Glycemic variability in individuals with type 2 diabetes mellitus in primary care measured by continuous glucose monitor device | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Valerija Lang, Principal Investigator — Association of teachers in general practice / family medicine
Locations (1):
- Association of teachers in general practice / family medicine, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baretic M, Bralic Lang V. Hypoglycemia in patients with type 2 diabetes treated with oral antihyperglycemic agents detected by continuous glucose monitoring: a multi-center prospective observational study in Croatia. BMC Endocr Disord. 2020 Mar 10;20(1):35. doi: 10.1186/s12902-020-0518-5. PMID 32151247